CLINICAL TRIAL: NCT03162289
Title: Intermittent Fasting Accompanying Chemotherapy in Gynecological Cancers - a Randomized, Controlled, Two-armed Intervention Study
Brief Title: Intermittent Fasting Accompanying Chemotherapy in Gynecological Cancers
Acronym: FIT2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FIT 2
Record Dates: First submitted 2017-05-10; First posted 2017-05-22 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Fasting; Vegan
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Fasting | interventions — Angptl4 protein, mouse; Diet, Vegan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting (Active Comparator): 60-72 h-modified fasting (36-48 h before and 24 h after chemotherapy)
  Interventions: Other: Fasting
- Vegan (Active Comparator): 60-72 h-vegan diet (36-48 h before and 24 h after chemotherapy)
  Interventions: Other: Vegan

INTERVENTIONS:
Other: Fasting — Patients follow a modified fasting regime of 60-72 h (36-48 h before and 24 h after CT) with a dietary energy supply of 350-400kcal per day with vegetable juices during the first four cycles of CT. During the rest of the CT cycles they will observe two days of caloric restriction (24 h before and after CT). Between CTs a mainly vegetarian diet will be performed and the patients are encouraged to follow a pattern of time restricted feeding with 14 h fasting over night at least for six days a week. The patients will receive an individual nutrition training by trained nutritionists.
  Arms: Fasting
Other: Vegan — Patients follow a 60-72 h vegan diet with sugar restriction (36-48 h before and 24 h after CT) during the first four cycles of CT. During the rest of the CT cycles they will observe two days of vegan and sugar-restricted diet (24 h before and after CT). Between CTs a mainly vegetarian diet will be performed. The patients will receive an individual nutrition training by trained nutritionists.
  Arms: Vegan

SUMMARY:
The aim of this trial is an evaluation of the effectiveness of intermittent fasting as a supplementary therapy in patients with breast cancer and ovarian cancer in respect to quality of life, reduction of side effects and possible reduction in tumor progression.

DETAILED DESCRIPTION:
Chemotherapy (CT) is a basic element in the therapy of gynecological oncologic diseases besides surgery, antibody therapy, anti-hormonal therapy and radiation. The chemotherapeutic intervention can be experienced physically and psychologically as a severe stress due to unwanted acute and also relevant long term side effects. It is even possible that because of severe side effects the CT can not be continued and main goals of the therapy like tumor reduction or elimination can not be achieved. Except of some medicinal approaches (such as antiemetics) or therapeutic exercise, not many therapeutic approaches are known to help reduce CT induced side effects. Against this background it is important to identify and scientifically evaluate new approaches to reduce the side effects of CT. The aim of this study is to verify the effectiveness of intermittent fasting as a potentially helpful supportive therapy in CT. In a prior pilot study of our institute with 34 breast- and ovarian cancer patients showed beneficial effects of an intermittent fasting of 72-84 h parallel to the application of the CT (manuscript submitted in Cancer Science).

The results of this confirmatory study are therefore of potentially high clinical relevance for all chemotherapeutically treated patients.

Long term goal: This study can lead to the improvement of tolerance and effectiveness of chemotherapeutic tumor therapy through accompanying intense nutritional therapy interventions. Beyond that it can be the starting point of a following multi-center randomized controlled study.

A large variety of animal experimental studies as well as three smaller pilot studies suggest that intermittent fasting can reduce the unwanted side effects of CT and enhance the quality of life. It is being speculated that the anti-tumor effect of fasting is enhanced through the reduction of the Insulin-like growth factor-1 (IGF-1) and mTOR as well as p53-signalling molecules (differential stress resistance).

But it is still unclear whether the possible beneficial effect that intermittent fasting shows can only be reached by subtotal caloric restriction or a significant reduction of the intake of animal proteins and refined sugar could also cause a similar decrease in IGF-1.

Against this background this confirmatory study aims to test the hypothesis that CT in the adjuvant and neoadjuvant treatment of breast- and ovarian cancer is better tolerable under intermittent fasting than under a normo-caloric vegan and sugar-reduced diet.

ELIGIBILITY:
Diagnosed, gynecological, malignant tumor disease (non-metastatic ovarian or breast cancer).

Other inclusion criteria:

* Age 18-75 years
* Cancer is treated conventionally with an adjuvant or neo-adjuvant protocol with at least 4 CT cycles

The following CTs are considered for breast carcinoma:

* - (EC, Sparano) 4 x Epirubicin and Cyclophosphamide, followed by 12 cycles Paclitaxel weekly
* - (AC, Henderson) 4 x Doxorubicin, cyclophosphamide, followed by 4 cycles Docetaxel every three weeks

If the recruitment rate is not reached, further CT protocols can be accepted.

CT for patients with ovarian cancer: According to current protocols, at least 4 planned cycles. For the study a maximum of 8 cycles are considered (except therapy with Taxol).

Exclusion Criteria:

* Reduction in CT dose compared to usual dosage
* Excessive underweight (BMI <19kg / m2) or actual weight reduction > 3kg or > 5kg in the last 1 or 3 months.
* Pre-existing eating disorder (Anorexia nervosa, Bulimia)
* Renal insufficiency (creatinine> 2mg / dl)
* Severe disease or other disease with a significant reduction in mobility and overall vitality
* Diabetes mellitus
* No inclusion in other study protocol
* Lack of email address and Internet access (due to electronic CRF)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
FACT-G | Date of inclusion (baseline), day -2 and +7 at each chemotherapy (CT) in triweekly cycles/-2 days at each CT in weekly cycles and +7 after the last weekly CT, 4 months after inclusion, 3 weeks after end of CT and 1, 2 and 3 years after inclusion
  Summarized change of FACT-G score

SECONDARY OUTCOMES:
Complete remissions | From date of randomization until the date of surgery
  Number of histologically proven complete remissions (ypT0ypN0 bzw. ypT0/is) after neoadjuvant CT
Millar Payne classification | after surgery/histological examination, an average 6 months after intervention start
  Histological classification according to Millar Payne scale

OTHER OUTCOMES:
Trial outcome index score (TOI) | Date of inclusion (baseline), day -2 and +7 at each chemotherapy (CT) in triweekly cycles/-2 days at each CT in weekly cycles and +7 after the last weekly CT, 4 months after inclusion, 3 weeks after end of CT and 1, 2 and 3 years after inclusion
  TOI
Total AC (FACT-B/FACT-O) | Date of inclusion (baseline), day -2 and +7 at each CT in triweekly cycles/-2 days at each CT in weekly cycles and +7 after the last weekly CT, 4 months after inclusion, 3 weeks after end of CT and 1, 2 and 3 years after inclusion
  According to kind of cancer (breast cancer/ ovarian cancer)
FACIT-F | Date of inclusion (baseline), day -2 and +7 at each CT in triweekly cycles/-2 days at each CT in weekly cycles and +7 after the last weekly CT, 4 months after inclusion, 3 weeks after end of CT and 1, 2 and 3 years after inclusion
  Fatigue
FACT-Tax,FACT/GynecologicOncologyGroup-Ntx | Date of inclusion (baseline), day -2 and +7 at each CT in triweekly cycles/-2 days at each CT in weekly cycles and +7 after the last weekly CT, 4 months after inclusion, 3 weeks after end of CT and 1, 2 and 3 years after inclusion
  Specific chemotherapy induced effects on quality of life and neurologic symptoms
Chemotherapy-Induced Peripheral Neuropathy Assessment Tool | Date of inclusion (baseline), day -2 and +7 at each CT in triweekly cycles/-2 days at each CT in weekly cycles and +7 after the last weekly CT, 4 months after inclusion, 3 weeks after end of CT and 1, 2 and 3 years after inclusion
  Chemotherapy-Induced Peripheral Neuropathy Assessment Tool
Hospital Anxiety and Depression Scale | Date of inclusion (baseline), day -2 and +7 at each CT in triweekly cycles/-2 days at each CT in weekly cycles and +7 after the last weekly CT, 4 months after inclusion, 3 weeks after end of CT and 1, 2 and 3 years after inclusion
  Hospital Anxiety and Depression Scale
Side effects of CT | Date of inclusion (baseline), day -2 and +7 at each CT in triweekly cycles/-2 days at each CT in weekly cycles and +7 after the last weekly CT, 4 months after inclusion, 3 weeks after end of CT and 1, 2 and 3 years after inclusion
  Likert scales
Weight | Timing varies according to individual therapy plan, Date of inclusion (baseline) and up to 3 years after inclusion
  Documentation according to the standard documentation rules of the German Tumour Centres Work Group, Weight in kilograms
BMI | Timing varies according to individual therapy plan, Date of inclusion (baseline) and up to 3 years after inclusion
  Documentation according to the standard documentation rules of the German Tumour Centres Work Group, BMI in kg/m^2
Blood panel | Timing varies according to individual therapy plan, Date of inclusion (baseline) and up to 3 years after inclusion
  Documentation according to the standard documentation rules of the German Tumour Centres Work Group, units auf measure according to SI units
Blood values for liver function | Timing varies according to individual therapy plan, Date of inclusion (baseline) and up to 3 years after inclusion
  Documentation according to the standard documentation rules of the German Tumour Centres Work Group, units auf measure according to SI units
Blood values for renal function (Krea, Hst.) | Timing varies according to individual therapy plan, Date of inclusion (baseline) and up to 3 years after inclusion
  Documentation according to the standard documentation rules of the German Tumour Centres Work Group, units auf measure according to SI units
IGF-1, Insulin, Blood glucose | Baseline, after 4 months and before each of the first 4 CTs meaning approx week 1,4,7 and 10 after intervention start
  Explorative measurements in blood samples in subgroup of 20 patients
Long-term explorative measurements: frequency of recurrence | 1, 2 and 3 years after baseline
  Information taken from the documentation of the treatment, visits and questionnaires
Long-term explorative measurements: e.g. polyneuropathy, cardiomyopathy | 1, 2 and 3 years after baseline
  Information taken from the documentation of the treatment, visits, questionnaires and interview
ketone bodies | Baseline, after 4 months and before each of the first 4 CTs meaning approx week 1,4,7 and 10 after intervention start
  Explorative measurements in capillary blood, only in subpopulation of n=20
Elective items of the "Common Terminology Criteria for Adverse Events (CTCAE) | Baseline, 3 weeks after end of CT, 1,2,3 years after baseline
  Elective items of the "Common Terminology Criteria for Adverse Events (CTCAE)"
Qualitative interviews in focus groups | Baseline, 6 months
  Qualitative interviews in focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Study Principal Investigator Charite
Locations (8):
- Germany (8):
  - Albert-Ludwigs-University of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg
  - Ernst-von-Bergmann Klinikum, Klinik für Gynäkologie und Geburtshilfe, Potsdam, Brandenburg
  - Brustzentrum Charite Campus Mitte, Berlin
  - Vivantes Brustzentrum, Berlin
  - Charité Virchow Klinikum, Berlin
  - Brustzentrum Krankenhaus Waldfriede, Berlin
  - Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus, Berlin

REFERENCES:
- [Derived] Koppold-Liebscher D, Kessler CS, Steckhan N, Bahr V, Kempter C, Wischnewsky M, Hubner M, Kunz B, Paul M, Zorn S, Sari S, Jeitler M, Stange R, Michalsen A. Short-term fasting accompanying chemotherapy as a supportive therapy in gynecological cancer: protocol for a multicenter randomized controlled clinical trial. Trials. 2020 Oct 15;21(1):854. doi: 10.1186/s13063-020-04700-9. PMID 33059765